CLINICAL TRIAL: NCT03746730
Title: ROLE OF Gray Scale and Doppler Ultrasound in Diagnosis of Parotid and Submandibular Gland Diseases
Brief Title: Role of US,Doppler in Major Salivary Gland Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, galal mohamed galal, Prinicible investigator, Assiut University
Other Study IDs: US,Doppler salivary diseases
Record Dates: First submitted 2018-09-30; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Salivary Gland Diseases
MeSH Terms: conditions — Salivary Gland Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasound — gray scale and doppler ultrasound

SUMMARY:
To evaluate the role of gray scale and Doppler ultrasound in characterizing of parotid and submandibular gland lesions in comparison to biopsy if needed

DETAILED DESCRIPTION:
* Salivary glands are affected by variety of disease processes which include infective, inflammatory, systemic, obstructive and neoplastic conditions . Clinical examination alone will not provide the correct diagnosis of salivary gland pathologies. Thus, radiological evaluation is essential in correct diagnosis .

USG plays a significant and crucial role in the diagnosis and management of salivary gland lesions. Results of the USG examination alone may suggest the final diagnosis or provide important differential diagnostic data . USG can differentiate intraglandular from extraglandular lesions in 98% of cases. It can differentiate salivary gland lesions as focal or diffuse. Characterisation of focal lesions into benign and malignant can be done by evaluation of edges. With high resolution transducers USG is better than CT or MRI in detection of unsharp borders .

Color Doppler findings are helpful in characterising the pathologies. It is helpful in diagnosing pleomorphic adenoma. Doppler findings of intralesional vascularity, type and grade of vascularity, PSV, RI and PI are useful in differentiating benign from malignant tumours . Pathological diagnosis can be established by Fine Needle Aspiration Cytology (FNAC). FNAC is preferably done under USG guidance. This helps in further enhancing ability of USG to differentiate between benign and malignant lesions .

Other radiological investigations for evaluation of salivary gland pathologies are plain radiography, sialography, CT, MRI and PET-CT .

Sometimes it is not possible to visualize lesions completely on USG because of their location, extension into the deep lobe of the parotid gland or behind the acoustic shadow of the mandible In these situations, further imaging with CT or MRI is necessary.

ELIGIBILITY:
Inclusion Criteria:

- Patients in different age and sex groups with neck swelling, pain or any complaint related to major salivary gland detected by clinical examination.

Exclusion Criteria:

* patients who refused to sign a consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients in different age and sex groups with neck swelling, pain or any complaint related to parotid and submandibular gland detected by clinical examination.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
the role of gray scale and Doppler ultrasound in characterizing of parotid and submandibular gland diseases in comparison to biopsy if needed | baseline
  the role of gray scale and Doppler ultrasound in characterizing of parotid and submandibular gland diseases in comparison to biopsy if needed

REFERENCES:
- [Background] Zhang W, Zuo Z, Luo N, Liu L, Jin G, Liu J, Su D. Non-enhanced MRI in combination with color Doppler flow imaging for improving diagnostic accuracy of parotid gland lesions. Eur Arch Otorhinolaryngol. 2018 Apr;275(4):987-995. doi: 10.1007/s00405-018-4895-6. Epub 2018 Feb 12. PMID 29430614
- [Background] Rzepakowska A, Osuch-Wojcikiewicz E, Sobol M, Cruz R, Sielska-Badurek E, Niemczyk K. The differential diagnosis of parotid gland tumors with high-resolution ultrasound in otolaryngological practice. Eur Arch Otorhinolaryngol. 2017 Aug;274(8):3231-3240. doi: 10.1007/s00405-017-4636-2. Epub 2017 Jun 13. PMID 28612315